CLINICAL TRIAL: NCT01531686
Title: An Observational Study to Determine the Safety and Effectiveness of Intraosseous Vascular Access for the Delivery of CT Contrast Dye
Brief Title: Observational Study of CT Dye Administration Through the Intraosseous Vascular Access Route
Status: Terminated | Type: Observational
Why Stopped: Slow rate of enrollment
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Organization: Teleflex (Industry)
Other Study IDs: 2011-02
Record Dates: First submitted 2012-02-03; First posted 2012-02-13 (Estimated); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2016-12

CONDITIONS: Patients With Intraosseous Vascular Access Requiring Computed Tomography (CT) Exam
Keywords: intraosseous vascular access; Computed Tomography (CT) examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intraosseous delivery of CT contrast dye — Delivery of CT contrast through intraosseous vascular access at the proximal humerus for CT examination.
  Other Names: EZ-IO

SUMMARY:
An observational study to determine the safety and effectiveness of Intraosseous (IO) vascular access for delivery of contrast dye for Computed Tomography (CT) examination. The hypothesis is that IO access can be safely and effectively used to deliver contrast medium for CT examination.

DETAILED DESCRIPTION:
An observational study to determine the safety and effectiveness of Proximal Humerus Intraosseous (IO) vascular access for delivery of contrast medium for Computed Tomography (CT) examination. The hypothesis is that Proximal Humerus IO access in conjunction with a pressure-limited power injection device can be safely and effectively used to deliver contrast medium for CT examination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Has received intraosseous (IO) vascular access at the proximal humerus insertion site via EZ-IO 45 mm needle set, as standard of care
* Requires Computed Tomography (CT) examination with contrast media delivery via proximal humerus intraosseous catheter, as standard of care
* Cognitively and physically able to give written consent to participate in the study or is obtained from a Legally Authorized Representative (LAR)

Exclusion Criteria:

* Fracture in target bone, or significant trauma to the site
* Excessive tissue and/or absence of adequate anatomical landmarks in target bone
* Infection in target area
* IO insertion in past 24 hours, prosthetic limb or joint or other significant orthopedic procedure in target bone
* Allergy to contrast media
* Imprisoned
* Pregnant
* Requires English language translation other than Spanish
* Has received proximal humerus IO access with an IO catheter other than the EZ-IO 45 millimeter (mm) needle set system
* Has existing proximal humerus IO access using the EZ-IO 45 mm needle set but IO catheter is mal-positioned or dislodged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have received proximal humerus intraosseous vascular access as standard of care via the EZ-IO 45 mm needle set and require Computed Tomography (CT) examination
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Philbeck, PhD, Study Director — Sponsor Company- Vidacare Corporation
Locations (4):
- United States (4):
  - Maricopa Medical Center, Phoenix, Arizona
  - Olive View UCLA Medical Center, Sylmar, California
  - Shands Critical Care Center and Cancer Hospital, Gainesville, Florida
  - Grand Strand Regional Medical, Myrtle Beach, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: observational study with patients enrolled in the emergency department
Groups:
- Proximal Humerus Intraosseous (IO) Computed Tomography (CT) Contrast: Adult patients in the emergency department receiving administration of contrast, via intraosseous (IO) vascular access established in the proximal humerus, for the purpose of computed tomography (CT) examination.
Period: Overall Study
Arm/Group | Proximal Humerus Intraosseous (IO) Computed Tomography (CT) Contrast
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Proximal Humerus Intraosseous (IO) Computed Tomography (CT) Contrast
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.25 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Adequacy of Computed Tomography (CT) Image
Description: Adequacy of CT image graded as adequate or inadequate indicating the ability to effectively administer the contrast medium needed for the indicated CT examination.
Time Frame: at time of CT examination average time is within 24 hours
Measure: Count of Participants; unit: Participants
Groups:
- Proximal Humerus Intraosseous (IO) Computed Tomography (CT) Contrast: Adult patients receiving administration of contrast for the purpose of computed tomography (CT) examination via intraosseous vascular access established in the proximal humerus, in the emergency department.
Arm/Group | Proximal Humerus Intraosseous (IO) Computed Tomography (CT) Contrast
Number analyzed (Participants) | 8
Participants
  CT Image graded as adequate | 7
  CT image graded as inadequate | 1

2. Primary Outcome: Incidence of Complication With Administration of Contrast for Computed Tomography (CT) Examination
Description: incidence of complications associated with the administration of contrast through the proximal humerus intraosseous (IO) route for CT examination
Time Frame: at time of CT examination average time is within 30 minutes
Measure: Number; unit: complications
Arm/Group | Proximal Humerus Intraosseous (IO) Computed Tomography (CT) Contrast
Number analyzed (Participants) | 8
complications | 1

ADVERSE EVENTS:
Time Frame: During the time of contrast administration until the end of follow up, up to 30 days
Description: patients were contacted 30 days following the contrast administration and asked if they experienced any adverse events. Per protocol, only other adverse events (not including serious adverse events) determined by the principal investigator (PI) to have at least a possible relationship to the contrast administration via the proximal humerus intraosseous vascular access route were recorded for this observational study by the PI.
Arm/Group | Proximal Humerus Intraosseous (IO) Computed Tomography (CT) Contrast
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less